CLINICAL TRIAL: NCT01832259
Title: A Neoadjuvant, Randomized, Phase II Study of Vascular Endothelial Growth Factor (VEGF) Tyrosine Kinase Inhibitor (Pazopanib) in Men With High-Risk Prostate Cancer Followed by Radical Prostatectomy and Pelvic Lymph Node Dissection
Brief Title: A Study of VEGF Tyrosine Kinase Inhibitor (Pazopanib) in Men With High-Risk Prostate Cancer Followed by Radical Prostatectomy and Pelvic Lymph Node Dissection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCI63129
Record Dates: First submitted 2013-03-21; First posted 2013-04-16 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Adenocarcinoma of the Prostate
MeSH Terms: interventions — pazopanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo arm (Placebo Comparator): Participants receiving placebo
  Interventions: Other: Placebo
- Pazopanib arm (Experimental): Participants receiving Pazopanib
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Pazopanib, 800 mg, orally daily for 28 days prior to radical prostatectomy.
  Arms: Pazopanib arm
Other: Placebo — Placebo tablet orally, daily for 28 days prior to radical prostatectomy.
  Arms: Placebo arm

SUMMARY:
The area around a tumor ("pre-metastatic niche") may be an area to which cancer cells are attracted. The study doctor will take blood and tumor samples to look for certain features linked with response to treatment so that they can predict which future patients may benefit from this therapy. The purpose of this study is to see if the drug pazopanib can be used to reduce the amount of pre-metastatic niche in the patient's lymph nodes (a common site for prostate cancer to spread). Down the line, this may help to prevent prostate cancer from coming back after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥ 18 years of age
* Histological documentation of adenocarcinoma of the prostate, with available biopsy pathology. Biopsy material must be available for pathologic review.
* All patients must meet one or more of the following disease features: clinical stage greater than or equal to T3; Primary Gleason score of 4 OR Gleason score of 8, 9 or 10; serum prostate-specific antigen (PSA) ≥ 20 ng/mL; Prostate MRI findings consistent with T3 disease; Any clinical stage and PSA (prostate-specific antigen) >10 and Gleason score 7; A Kattan nomogram predicted probability of being free from biochemical progression at 5 years after surgery of < 60%.
* Patients must have a PSA (prostate-specific antigen) ≥ 2 ng/mL at the time of diagnosis of prostate cancer or later.
* No prior radiation or chemotherapy for prostate cancer treatment.
* Scheduled for radical prostatectomy surgery.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Patients may have been treated with up to 4 months of androgen deprivation therapy.
* No clinical evidence of metastatic prostate cancer, or enlarged pelvic lymph nodes in the imaging studies.
* Resected lymph nodes must be provided for all subjects for biomarker analysis immediately (same day) after surgery (radical prostatectomy).
* Adequate organ system function as defined by study Protocol

  1. Subjects may not have had a transfusion within 7 days of screening assessment.
  2. Concomitant elevations in bilirubin and aspartate aminotransferase (AST)/alanine aminotransferase (ALT) above 1.0 x upper limit of normal (ULN) are not permitted.
  3. If urine protein count (UPC) =>1, then a 24-hour urine protein must be assessed. Subjects must have a 24-hour urine protein value <1 to be eligible.
* Subjects must provide written informed consent within one month prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow up.

Exclusion Criteria:

* Clinical evidence of metastatic prostate cancer.
* Prior malignancy. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years.
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to: Active peptic ulcer disease Known intraluminal metastatic lesion/s with risk of bleeding Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment.
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

  * Malabsorption syndrome or
  * Major resection of the stomach or small bowel.
* Corrected QT interval (QTc) > 480 msecs Note: Correction method should be reported
* History of any one or more of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft surgery
  * Symptomatic peripheral vascular disease
  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* No evidence of preexisting uncontrolled hypertension. If the patient has a history of elevated blood pressure at baseline then they must have controlled hypertension documented and confirmed by 2 consecutive blood pressure readings taken within 1 hour. The baseline systolic blood pressure readings must be =<140 mm Hg, and the baseline diastolic blood pressure readings must be =<90 mm Hg.

Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. Following antihypertensive medication initiation or adjustment, blood pressure (BP) must be re-assessed three times at approximately 2-minute intervals. At least 24 hours must have elapsed between anti-hypertensive medication initiation or adjustment and Blood Pressure measurement. These three values should be averaged to obtain the mean diastolic blood pressure (DBP) and the mean systolic blood pressure (SBP). The mean SBP / DBP ratio must be <140/90 mm Hg (OR 150/90 mm Hg, if this criterion is approved by the Huntsman Cancer Institute (HCI) Data Safety and Monitoring Committee (DSMC) Chair or Co-chair) in order for a subject to be eligible for the study (see protocol for details on Blood Pressure control and re-assessment prior to study enrollment).

* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major surgery).
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage Note: Lesions infiltrating major pulmonary vessels (contiguous tumour and vessels) are excluded; however, the presence of a tumor that is touching, but not infiltrating (abutting) the vessels is acceptable (CT (computed tomography) with contrast is strongly recommended to evaluate such lesions).

  * Large protruding endobronchial lesions in the main or lobar bronchi are excluded; however, endobronchial lesions in the segmented bronchi are allowed.
  * Lesions extensively infiltrating the main or lobar bronchi are excluded; however, minor infiltrations in the wall of the bronchi are allowed.
* Recent hemoptysis (=> ½ teaspoon of red blood within 8 weeks before first dose of study drug).
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Unable or unwilling to discontinue use of prohibited medications listed in the protocol for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.
* Treatment with any of the following anti-cancer therapies:

  * radiation therapy, chemotherapy, immunotherapy, biologic therapy, investigational therapy
  * surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of Pazopanib
* Administration of any non-oncologic investigational drug within 30 days or 5 half lives whichever is longer prior to receiving the first
* Any ongoing toxicity from prior hormonal therapy that is >Grade 1 and/or that is progressing in severity.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2017-02-07 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Agarwal, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Maughan BL, Pal SK, Gill D, Boucher K, Martin C, Salgia M, Nussenzveig R, Liu T, Hawks JL, Batten J, Nachaegari G, Stephenson R, Lowrance W, Jones J, Dechet C, Agarwal N. Modulation of Premetastatic Niche by the Vascular Endothelial Growth Factor Receptor Tyrosine Kinase Inhibitor Pazopanib in Localized High-Risk Prostate Cancer Followed by Radical Prostatectomy: A Phase II Randomized Trial. Oncologist. 2018 Dec;23(12):1413-e151. doi: 10.1634/theoncologist.2018-0652. Epub 2018 Nov 1. PMID 30575560

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Arm | Pazopanib Arm
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Arm | Pazopanib Arm | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.33 (4.71) | 64.13 (6.26) | 63.73 (5.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Vascular Endothelial Growth Factor Receptor 1 (VEGFR1)-Positive Clusters
Description: Patients with high-risk, localized prostate cancer were treated with 28 days of Pazopanib or placebo, after which they underwent radical prostatectomy. During prostatectomy, benign pelvic lymph node tissue was collected and subsequently analyzed for the average number of VEGFR1-positive clusters in 8 distinct 40x microscopic fields as an indicator of pre-metastatic niche formation.
Time Frame: 1 month
Population: The tissue of one patient on the Pazopanib arm and two patients on the Placebo arm was not able to be analyzed. Another patient on the Pazopanib arm had surgery delayed by a few weeks following stopping study medication and was determined to be unevaluable, resulting in 13 patients analyzed on each arm.
Measure: Mean (Standard Deviation); unit: VEGFR1+ clusters per hpf
Arm/Group | Placebo Arm | Pazopanib Arm
Number analyzed (Participants) | 13 | 13
VEGFR1+ clusters per hpf | 0.251560 (0.093458902) | 0.269518 (0.120773334)
Statistical Analysis 1: Comparison: Placebo Arm vs Pazopanib Arm; Test type: Superiority; p = 0.345, t-test, 1 sided

2. Secondary Outcome: Participants Experiencing Adverse Events
Description: Adverse events were assessed using the Common Terminology for Adverse Events (CTCAE) version 4. Each event was assigned a grade (1-5), with lower grades indicating milder events. All adverse events were recorded, regardless of attribution to study treatment. For a full listing of Adverse Events, please see the Adverse Events section of the Results for this study.
Time Frame: From first dose of study treatment to one month post-prostatectomy (approximately 2 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Arm | Pazopanib Arm
Number analyzed (Participants) | 15 | 15
Participants
  Participants experiencing Grade 1-2 Adverse Events | 15 | 15
  Participants experiencing Grade 3-4 Adverse Events | 0 | 4

3. Secondary Outcome: Biochemical Recurrence Progression Free Survival Rate
Description: Following prostatectomy, patients' Prostate Specific Antigen (PSA) lab values were collected for up to two years. Biochemical recurrence was defined as the first PSA lab value of greater than or equal to 0.2 ng/mL following prostatectomy. Biochemical recurrence progression free survival rate was defined as the percent chance of 1 year survival with no biochemical recurrence.
Time Frame: 2 years
Population: Two patients on the Pazopanib arm were not evaluable, one due to prostatectomy not being completed, and one due to prostatectomy being delayed outside of protocol windows.
Measure: Number (95% Confidence Interval); unit: percent chance of survival
Arm/Group | Placebo Arm | Pazopanib Arm
Number analyzed (Participants) | 15 | 13
percent chance of survival | 73.3 [54.0 to 99.5] | 92.3 [78.9 to 100]
Statistical Analysis 1: Comparison: Placebo Arm vs Pazopanib Arm; Test type: Superiority; p = 0.46, Log Rank

ADVERSE EVENTS:
Time Frame: Adverse events were collected for approximately 2 months (from first dose of study medication to 1 month post-prostatectomy).
Description: The occurrence of adverse events was sought by non-directive questioning of the patient at each visit or phone contact during the study. Adverse events were also detected when they were volunteered by the patient during or between visits or through physical examination, laboratory test, or other assessments.
Arm/Group | Placebo Arm | Pazopanib Arm
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=15) | Pazopanib Arm (N=15)
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Agitation (Psychiatric disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 4 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bladder spasm (Renal and urinary disorders) | 2 | 0
Bloating (Gastrointestinal disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (2) | 1
Burn (Injury, poisoning and procedural complications) | 1 | 0
Irregular heartbeat (Cardiac disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 (4) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Creatinine increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 5 (6) | 6
Dizziness (Nervous system disorders) | 2 | 3
Dry mouth (Gastrointestinal disorders) | 1 (2) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 2 (3) | 2
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 0
Eye disorders - Other (Eye disorders) | 0 | 3
Fatigue (General disorders) | 6 | 9
Fever (General disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Flu like symptoms (General disorders) | 3 (4) | 1
Flushing (Vascular disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Loose stool (Gastrointestinal disorders) | 1 | 0
Generalized discomfort (General disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Genital edema (Reproductive system and breast disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 1
Hematoma (Vascular disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 2 | 1
Hemoglobin increased (Investigations) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Hot flashes (Vascular disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 (5) | 8 (12)
Hypotension (Vascular disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Localized edema (General disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (2)
Nausea (Gastrointestinal disorders) | 4 | 5 (6)
Oral dysesthesia (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 (3)
Pelvic pain (Reproductive system and breast disorders) | 1 | 2
Perineal pain (Reproductive system and breast disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
Phlebitis (Vascular disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 1
Hair color change (Skin and subcutaneous tissue disorders) | 0 | 3
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 3 (4)
Urinary incontinence (Renal and urinary disorders) | 4 | 2
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT01832259/Prot_SAP_000.pdf